CLINICAL TRIAL: NCT03371511
Title: Sources of Bacterial Contamination in Human Milk Samples From the Milk in Life Conditions (MiLC) Trial
Brief Title: Sources of Bacterial Contamination in Human Milk Samples From the MiLC Trial
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Idaho (Other)
Responsible Party: Sponsor
Other Study IDs: 1608006566; 2T32DK007158-42 (NIH)
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Bacterial Communities
Keywords: Microbiota; Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Swabs were taken of women's dominant hand, the breast from which she donated milk (nipple, areola), their milk collection kit (bottle and flange), their pump (pump port and tubing), and their babies' mouths.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MiLC Cohort: Participants donated HM from two consecutive pumping sessions at home. Women pumped once with their own pump and milk collection kit, and once with a sterile and sterile collection kit. Both pumping sessions occurred at participants' homes between 0700 and 1100 hours. The second pumping session occurred within 3 hr (+/- 30 min) after the beginning of the first. Randomization was used to determine which pump was used first. Women elected from which breast they donated their HM and were asked not to nurse on that side 2 hr before the first pumping session and not until after the second. Before women pumped with their own pump, swabs were taken of the breast from which HM was donated, the women's dominant hand, their own bottle/flange, their own pumps (port of pump and tubing), and their babies' mouths.
  There was only one group but stratified enrollment was used to ensure equal numbers of women whose infants consumed HM only and women whose infants consumed HM and complementary foods.

SUMMARY:
This observational study is a sub-study of the MiLC Trial (ClinicalTrials.gov Identifier: NCT03123874). Our objective is to characterize the bacterial communities of women's breasts, hands, their pump and milk collection kit, and their babies' mouths among the participants of the MiLC Trial. As part of the original protocol, we collected swabs of each of these areas from each dyad before women pumped with their own pumps. By characterizing these communities, we can identify from where the bacteria in human milk (HM) originates, and determine whether pumping with mother's own pumps enriches the bacterial communities of HM compared to pumping with a sterile pump.

ELIGIBILITY:
Inclusion Criteria:

* Mother-infant dyads who participated in the MiLC Trial.

Exclusion Criteria:

* Anyone who did not participate in the MiLC Trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Lactating women
Study Population: Mother-infant dyads who participated in the MiLC Trial. These were healthy, lactating women 18 years or older. Women had no signs of breast infection and self-reported that they nor their infants had signs/symptoms of acute illness 7 days before participating in the study. We also restricted participation to women who pumped with electric breast pumps, who could donate 1 oz of their milk on two consecutive pumping sessions from the same breast, and women whose infants had not consumed formula within the past 2 weeks. A full description of eligibility criteria can be found on the original protocol (ClinicalTrials.gov Identifier: NCT03123874).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-03 (Actual)

PRIMARY OUTCOMES:
Bacterial communities | 0 days after pumping
  Bacterial communities of each swab (breast, hand, mother's own bottle/flange, mother's own pump/tubing, and infant mouth) will be determined by next-generation sequencing of the V1-V3 region of the 16S rRNA bacterial gene.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Reyes, MS, Study Director — Cornell University; Kathleen M Rasmussen, ScD, Principal Investigator — Cornell University; Anthony G Hay, PhD, Principal Investigator — Cornell University
Locations (1):
- Hay Laboratory, B75C Wing Hall, Cornell University, Ithaca, New York, United States